CLINICAL TRIAL: NCT00930891
Title: Randomized Phase II-III Study of Bevacizumab 7,5 mg/kg in Combination With Chemotherapy Versus Chemotherapy in Extensive-Disease Small-Cell Lung Cancer After Response to Chemotherapy : PCDE (cisPlatin - Cyclophosphamide - epiDoxorubicin - Etoposide) or PE (cisPlatin - Etoposide)
Brief Title: Bevacizumab in Extensive Small Cell Lung Cancer
Acronym: CPC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0802; 2009-010187-42
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Small Cell Lung Cancer
Keywords: Extensive-Disease Small-Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — 2,2',4,4',5-pentachlorodiphenyl ether; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): 4 additional cycles of chemotherapy
  Interventions: Drug: Standard Chemotherapy (PCDE or PE); Drug: Prerandomization Chemotherapy (PCDE or PE)
- Arm B (Experimental): 4 additional cycles of chemotherapy + bevacizumab
  Interventions: Drug: Experimental Treatment (PCDE or PE + bevacizumab); Drug: Prerandomization Chemotherapy (PCDE or PE)

INTERVENTIONS:
Drug: Standard Chemotherapy (PCDE or PE) — PCDE: cisPlatin 75 mg/m² D2 ; Cyclophosphamide 300 mg/m² D1 to D3; 4'-epiDoxorubicin 30 mg/m² D1; Etoposide 75 mg/m² D1 to D3, 4 cycles
  PE: cisPlatin 80 mg/m², D2; Etoposide 120 mg/m² D1 to D3, 4 cycles
  Arms: Arm A
Drug: Experimental Treatment (PCDE or PE + bevacizumab) — PCDE: cisPlatin 75 mg/m² D2; Cyclophosphamide 300 mg/m² D1 to D3; 4'-epiDoxorubicin 30 mg/m² D1; Etoposide 75 mg/m² D1 to D3, 4 cycles Bevacizumab 7.5 mg/kg, D1, until progression
  PE: cisPlatin 80 mg/m², D2; Etoposide 120 mg/m² D1 to D3, 4 cycles Bevacizumab 7.5 mg/kg, D1, until progression
  Arms: Arm B
Drug: Prerandomization Chemotherapy (PCDE or PE) — PCDE: cisPlatin 75 mg/m² D2; Cyclophosphamide 300 mg/m² D1 to D3; 4'-epiDoxorubicin 30 mg/m² D1; Etoposide 75 mg/m² D1 to D3, 2 cycles
  PE: cisplatin 80 mg/m², D2; Etoposide 120 mg/m² D1 to D3, 2 cycles

SUMMARY:
Despite the fact that a substantial response rate may be obtained in small-cell lung cancers (using double-drug chemotherapy: cisplatin-etoposide, PE), a cure remains an exception. More aggressive regimens remain controversial and recent attempts at increasing dose-intensity have been restricted to patients with a more favourable presentation.

Bevacizumab is a humanized monoclonal antibody which binds to VEGF (Vascular Endothelial Growth Factor). In association with double-drug standard chemotherapies, it has been proven that bevacizumab can improve survival of previously untreated advanced non-small-cell lung cancers (NSCLC), compared to chemotherapy without bevacizumab). Such promising effects on NSCLC deserve to be tested on small-cell lung cancers.

In this trial (IFCT-0802), standard chemotherapy (PCDE or PE) will be compared to experimental treatment (PCDE or PE + bevacizumab 7.5 mg/kg) for previously untreated SCLC patients.

ELIGIBILITY:
Inclusion Criteria (must be checked at the inclusion, week -8):

* Small-Cell Lung Cancer histologically or cytologically proved
* Extended disease as defined by Veteran's Administration Lung Cancer Group (VALG)
* At least one unidimensionally measurable lesion (RECIST criterion)
* Age between 18 and 75 years
* Weight loss < 10% for the last three month
* Performance Status (PS)≤ 2
* Creatininemia < 110 µmol/L and creatinin clearance > 60 mL/min
* Neutrophils ≥ 1,500/µL and platelets ≥ 100,000/µL
* Bilirubin ≤ 1.5 x normal value
* Transaminases, Alkaline Phosphatase ≤ 2.5 x ULN excepted in case of liver metastasis (5xULN)
* Left ventricular ejection fraction (measured by echocardiographic or isotopic method) > 50% if PCDE is planned
* Electrocardiogram without uncontrolled coronaropathy
* Signed informed consent

Randomization Criteria (to be checked during the randomization (week 0)):

* Partial or complete tumoral response as defined by RECIST
* All chemotherapy-induced toxicities decreased to level ≤ 2 as defined by NCI CTC VS 3 (except for alopecia)
* Inclusion criteria concerning creatininemia, clearance, neutrophils, platelets, transaminases, alkaline phosphatases and left ventricular ejection fraction must be checked again

Exclusion Criteria:

* Non-Small-Cell Lung Cancer or mixed cancer (small-cell / non-small-cell)
* Previous antitumoral treatment of the small-cell lung cancer (chemotherapy, radiotherapy, immunotherapy, surgery)
* Non-extended disease as defined by VALG
* Natremia < 125 mmol/L
* Hypercalcemia whereas a corrective treatment
* Pathology contra-indicating the hyper-hydration
* Hemoptysis in the last three months
* Tumor invading large vessels or invading the proximal trachea-bronchial tree (visible at the medical imagery). Investigator or radiologist must reject tumors adjoining, merging or extending to large vessel's lumen (for example : pulmonary artery, superior vena cava)
* Symptomatic cerebral or meningeal metastasis
* Other cancer in progress or medical history of cancer in the five last years (excepted basal cell carcinoma or in situ cervical cancer of the uterus.
* Important surgical intervention (including surgical biopsy), traumatic lesion during 28 days before starting the treatment, or anticipation of an important surgical intervention during the study
* Minor surgical intervention, including implanting permanent catheter during the 24 hours before the first administration of bevacizumab
* Unhealed wound, evolutive gastroduodenal ulcer, fractured bone
* Medical history of abdominal fistula, trachea-oesophageal fistula, of another type with a severity rank of 4, gastrointestinal perforation or intraabdominal abscess during 6 month before inclusion
* Ongoing or recent use of aspirin (during 10 days before the first administration of bevacizumab) (>325 mg/day) or use of another platelet aggregation inhibitor (dipyridamole, ticlopidine, clopidogrel > 75 mg/day), or ongoing or recent use of a therapeutic dose (during 10 days before the first administration of bevacizumab) of anticoagulant or thrombolytic drugs per os or in parenteral injection. Prophylactic use of anticoagulant drug is allowed
* Medical history or genetic predisposition to bleeding or coagulopathy
* Clinically significative cardiac disease: infarct or CVA during 6 month before inclusion, unstable angina, congestive cardiac failure level > II as defined by New York Heart Association (NYHA) or cardiac arrythmia needing a specific treatment which risk to interfere with the study, or uncontrolled arrythmia.
* Known allergy or hypersensibility to monoclonal antibodies (bevacizumab), to chinese hamster ovary cells or to any humanized or recombinant antibody
* Uncontrolled high blood pressure (systolic pressure > 150 mm Hg and/or diastolic pressure > 100 mm Hg), with or without hypotension treatment. Patients presenting an high blood pressure are eligibles if their treatment can decrease their blood pressure to the values required by the protocol.
* Severe ongoing infectious disease or fever > 38.5°C or evidence of any other pathology, organic or neurologic functions deterioration, physical examination or laboratory result which cause suspicion of a disease which contra-indicate use of any studied treatment.
* Woman with a positive pregnancy test or who has not made a pregnancy test (unless pregnancy risk can be excluded)
* Lactating woman
* Sexually active woman who don't use hormonal or mechanical contraceptive method or sexually active man who has a sexually active partner who don't want to use an effective contraceptive method during the course of the study and during the 6 months after last treatment administration
* Patient who as already been included and treated in the present study
* Patient who participate or who has participated in another study during 4 weeks before treatment administration
* Patient who receive a previous antiangiogenic treatment (experimental or commercial : bevacizumab, thalidomide, CP-547632, sunitinib, sorafenib...)
* Geographical or psychological condition which not allowed a good comprehension or compliance to protocol
* Liberty deprived patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response + partial response) | 6 weeks after randomization

SECONDARY OUTCOMES:
Progression-free survival | 12 weeks
Complete response length | 12 weeks
Quality of life | 12 weeks
Toxicities | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PUJOL, Pr, Principal Investigator — CHRU Montpellier
Locations (60):
- France (60):
  - Annemasse - CH, Ambilly
  - Angers - CHU, Angers
  - Armentières - CH, Armentières
  - CHU Besancon - Pneumologie, Besançon
  - Centre F. Baclesse, Caen
  - CHU - Pneumologie, Caen
  - Cahors - CH, Cahors
  - Chauny - CH, Chauny
  - Chalons-en-Champagne - CH, Châlons-en-Champagne
  - Hôpital Percy-Armées - Pneumologie, Clamart
  - Clermont Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - CH - Compiègne, Compiègne
  - Créteil - CHI, Créteil
  - Dijon - CAC, Dijon
  - Dijon - CHU, Dijon
  - Draguignan - CH, Draguignan
  - CHU Grenoble - pneumologie, Grenoble
  - Harfleur - Clinique du Petit Colmoulins, Harfleur
  - Saint Omer - CHI, Helfaut
  - Jonzac - CH, Jonzac
  - Chartres - CH, Le Coudray
  - Centre Hospitalier - Pneumologie, Le Mans
  - CH, Longjumeau
  - APHM - Hôpital Sainte Marguerite, Marseille
  - Marseille - CRLCC, Marseille
  - Maubeuge - Polyclinique du Parc, Maubeuge
  - Meaux - CH, Meaux
  - Metz - CHR, Metz
  - Mont de Marsan - CH, Mont-de-Marsan
  - Montpellier - CHRU, Montpellier
  - Mulhouse - CH, Mulhouse
  - Neuilly - Hôpital Américain de Paris, Neuilly
  - Nevers - CH, Nevers
  - Nice - CAC, Nice
  - Orléans - CH, Orléans
  - APHP - Saint-Antoine - pneumologie, Paris
  - APHP - Hopital Tenon - Pneumologie, Paris
  - Pau - CH, Pau
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - Reims - CHU, Reims
  - Reims - CRLCC, Reims
  - Rouen - CHU, Rouen
  - Saint Brieuc - CHG, Saint-Brieuc
  - Saint Nazaire - Centre Etienne Dolet, Saint-Nazaire
  - Saint Priest en Jarez - ICL, Saint-Priest-en-Jarez
  - Saint Quentin - CH, Saint-Quentin
  - Saverne - CH, Saverne
  - Senlis - CH, Senlis
  - Nouvel Hopital Civil - Pneumologie, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Thonon les bains, Thonon-les-Bains
  - Toulon - HIA, Toulon
  - CHU Toulouse - Pneumologie, Toulouse
  - Toulouse - Clinique Pasteur, Toulouse
  - Tours - CHU, Tours
  - Nancy - CHU, Vandœuvre-lès-Nancy
  - Verdun - CHG, Verdun
  - Vesoul - CHI, Vesoul
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Pujol JL, Breton JL, Gervais R, Tanguy ML, Quoix E, David P, Janicot H, Westeel V, Gameroff S, Geneve J, Maraninchi D. Phase III double-blind, placebo-controlled study of thalidomide in extensive-disease small-cell lung cancer after response to chemotherapy: an intergroup study FNCLCC cleo04 IFCT 00-01. J Clin Oncol. 2007 Sep 1;25(25):3945-51. doi: 10.1200/JCO.2007.11.8109. PMID 17761978
- [Background] Pujol JL, Daures JP, Riviere A, Quoix E, Westeel V, Quantin X, Breton JL, Lemarie E, Poudenx M, Milleron B, Moro D, Debieuvre D, Le Chevalier T. Etoposide plus cisplatin with or without the combination of 4'-epidoxorubicin plus cyclophosphamide in treatment of extensive small-cell lung cancer: a French Federation of Cancer Institutes multicenter phase III randomized study. J Natl Cancer Inst. 2001 Feb 21;93(4):300-8. doi: 10.1093/jnci/93.4.300. PMID 11181777
- [Background] Horn L, Dahlberg SE, Sandler AB, Dowlati A, Moore DF, Murren JR, Schiller JH. Phase II study of cisplatin plus etoposide and bevacizumab for previously untreated, extensive-stage small-cell lung cancer: Eastern Cooperative Oncology Group Study E3501. J Clin Oncol. 2009 Dec 10;27(35):6006-11. doi: 10.1200/JCO.2009.23.7545. Epub 2009 Oct 13. PMID 19826110
- [Result] Pujol JL, Lavole A, Quoix E, Molinier O, Souquet PJ, Barlesi F, Le Caer H, Moro-Sibilot D, Fournel P, Oster JP, Chatellain P, Barre P, Jeannin G, Mourlanette P, Derollez M, Herman D, Renault A, Dayen C, Lamy PJ, Langlais A, Morin F, Zalcman G; French Cooperative Thoracic Intergroup (IFCT). Randomized phase II-III study of bevacizumab in combination with chemotherapy in previously untreated extensive small-cell lung cancer: results from the IFCT-0802 trialdagger. Ann Oncol. 2015 May;26(5):908-914. doi: 10.1093/annonc/mdv065. Epub 2015 Feb 16. PMID 25688059
- [Derived] Negre E, Coffy A, Langlais A, Daures JP, Lavole A, Quoix E, Molinier O, Greillier L, Audigier-Valette C, Moro-Sibilot D, Westeel V, Morin F, Roch B, Pujol JL. Development and Validation of a Simplified Prognostic Score in SCLC. JTO Clin Res Rep. 2020 Feb 12;1(1):100016. doi: 10.1016/j.jtocrr.2020.100016. eCollection 2020 Mar. PMID 34589918
- See also: IFCT official website — http://www.ifct.fr